CLINICAL TRIAL: NCT03338634
Title: Pilot Testing of Food Images in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Assistant Professor, Department of Nutritional Sciences and Food Science, Penn State University
Other Study IDs: Pilot Food Images
Record Dates: First submitted 2017-10-11; First posted 2017-11-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Childhood Obesity; fMRI
Keywords: Portion Size Effect; Childhood Obesity; fMRI
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children 6 to 10: Children must be between the ages of 6-10 years-old at the time they participate. All children will be physically healthy and without diagnosed learning disorders. A parent or legal guardian must be able to accompany the child.

SUMMARY:
This is a single, un-replicated visit to the Children's Metabolic Kitchen and Eating Behavior Lab designed to gather data on children's responses to images used in MRI studies. Additionally, a demographic questionnaire for parents will be piloted.

DETAILED DESCRIPTION:
The Pilot Test Session will take place in the Children's Metabolic Kitchen and Eating Behavior Lab in Chandlee Laboratory. Up to four hundred subjects (200 children and 200 parents) may be recruited.

Child Procedures: Both Child and parent's current height and weight will be obtained. After being seated at a computer, they will complete the Children's Anxiety Meter-State (CAMS) and a Freddy Fullness pictorial hunger score. Then their ability to discriminate between portion sizes will be assessed. They will be shown several pictures of macaroni and cheese on a standard white plate with a grey tablecloth background and asked to determine which picture had a larger amount of food. Finally, they will view 180 pictures of common foods and non-food objects (office supplies). After each picture, children will be instructed to answer questions about the image (what is this image, how happy does it make you feel and how excited does it make you feel). Children will then score their hunger again with a Freddy Fullness pictorial hunger score and take a Post-Scanning Questionnaire.

Parent Procedures: Parent's current height and weight will be obtained and he/she will complete a demographic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Child is 6 to 10 years old
* Child is physically healthy and does not have a diagnosed learning disorder

Exclusion Criteria:

* Child is < 6 or > 10 years old
* Child is not physically healthy or has a diagnosed learning disorder

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents and their 6-10 year old children in Centre County, Pennsylvania and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Pilot Image Description by Children | baseline
  Once the child is comfortable in our lab and consent has been received, they will be shown a total of 150 - 200 pictures of foods and non-food objects (e.g. office supplies). They will also be shown control images that are blurred or scrambled versions of the test images. After each picture, children will be instructed answer questions about the image (ex. what is this image, how much do you like it, how large is it, etc.)

SECONDARY OUTCOMES:
Anthropometric Measures:weight | baseline
  The parent and child will be weighed in kg.
Anthropometric Measures:height | baseline
  The height of the parent and child will be measured in meters.
Demographic Questionnaire | baseline
  The parent will complete a fill-in the blank and multiple choice demographic questionnaire. No scales are used.
Freddy Fullness Scale Rating | baseline
  The child will complete a pictorial scale of fullness using a Freddy Scale. This is basically a vertical slider scale, with an empty stomach equaling 0 mm and a full stomach being 150 mm.
CAMS anxiety scale Rating | baseline
  The child will complete a CAMS anxiety scale questionnaire before viewing the images. This scale resembles a sliding scale thermometer. When the thermometer is empty, at zero, the child is calm and not nervous or worried. When the thermometer is full, the child is very, very nervous or worried.

OTHER OUTCOMES:
Post-Scanning Questionnaire | baseline
  After viewing the images and answering questions, children will be interviewed by the researcher to find out if they liked the procedure and whether or not they would refer their friends (to determine if other children are likely to enjoy the experience). There is no scale, the questions require a verbal answer.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Metabolic Kitchen and Children's Eating Behavior Lab, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared with other investigators by special request made by email to the PI (Kathleen L. Keller klk37@psu.edu). For investigators who request use of the data, we will request acknowledgement of our research group and Penn State University in any public presentation of the results obtained from this study.

REFERENCES:
- [Background] Burger KS, Stice E. Variability in reward responsivity and obesity: evidence from brain imaging studies. Curr Drug Abuse Rev. 2011 Sep;4(3):182-9. doi: 10.2174/1874473711104030182. PMID 21999692
- [Background] Bruce AS, Martin LE, Savage CR. Neural correlates of pediatric obesity. Prev Med. 2011 Jun;52 Suppl 1:S29-35. doi: 10.1016/j.ypmed.2011.01.018. Epub 2011 Feb 1. PMID 21291906
- [Background] De Silva A, Salem V, Matthews PM, Dhillo WS. The use of functional MRI to study appetite control in the CNS. Exp Diabetes Res. 2012;2012:764017. doi: 10.1155/2012/764017. Epub 2012 May 8. PMID 22719753
- See also: Dr. Kathleen Keller's current research — http://nutrition.hhdev.psu.edu/childrens-eating-lab